CLINICAL TRIAL: NCT06465160
Title: A Phase Ib, Open Label, Single or Repeated Dose Exploration Clinical Study to Evaluate the Safety and Therapeutic Effects of Infusion of MNV-201 (Autologous CD34+ Cells Enriched With Allogenic Placenta Derived Mitochondria) in Patients With Low-Risk Myelodysplastic Syndrome
Brief Title: A Study to Evaluate the MNV-201 in Patients With Low Risk MDS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Minovia Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNV-012
Record Dates: First submitted 2024-06-02; First posted 2024-06-18 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: Low Risk MDS; Anemia; Mitochondrial; Cell Therapy
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia

STUDY DESIGN:
Intervention Model Description: The study will have two parts: a single dose arm (Part 1) and a repeat dose arm (Part 2).
  Part 2 of the study will be subject to FDA's approval of individual patient re-dosing, after submission of patient-specific data to the FDA for review.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CD34+ cells enriched with allogenic placenta-derived mitochondria (Experimental): Participants will receive a single or repeated dose of MNV-201 product by Infusion after 5 days of mobilization by G-CSF and an apheresis procedure.
  Interventions: Biological: MNV-201 (Autologous CD34+ Cells Enriched with allogenic Placenta Derived Mitochondria)

INTERVENTIONS:
Biological: MNV-201 (Autologous CD34+ Cells Enriched with allogenic Placenta Derived Mitochondria) — The participant will undergo 5 days of mobilization by G-CSF administration (Neupogen) once a day during 5 days.
  On the 5th day, and after receiving the last dose of Neupogen, the participant will undergo Apheresis to collect CD34+ cells.
  MNV-201 consists of autologous CD34+ cells enriched with allogeneic placenta derived mitochondria. Autologous CD34+ cells are isolated from the participant's peripheral blood after mobilization by apheresis. Allogeneic mitochondria are isolated under aseptic conditions from healthy donor placenta, cryopreserved and qualified before use.
  Each product package will consist of a ready-for-injection sterile infusion bag containing clinical grade MNV-201 product for IV infusion for a single specified (autologous) participant.

SUMMARY:
Myelodysplastic syndromes (MDS) are a group of bone marrow failures that occur when the blood-forming cells in the bone marrow become abnormal leading to an abnormal differentiation and production of one or more blood cell types. According to the American Cancer Society, in the United States, MDS occurs at a rate of 4.8 cases for every 100,000 people; MDS affects an estimated 60,000 persons in the United States, with 10,000-15,000 new cases recorded each year. MDS is defined by ineffective haematopoiesis resulting in blood cytopenias (a reduction in the number of mature blood cells), and clonal instability with a risk of evolution to acute myeloid leukaemia (AML). Patients with MDS collectively have a high symptom burden and are also at risk of death from complications of cytopenias and AML. MDS is generally a disease that develops with ageing; the median age at diagnosis of MDS is ~70 years, and patients frequently have comorbid conditions. The goals of therapy for patients with MDS are to reduce disease-associated symptoms and the risk of disease progression and death, thereby improving both quality and quantity of life.

Minovia Therapeutics Ltd. ("Minovia") is a biotech company developing novel therapeutics based on its mitochondrial augmentation technology (MAT). MNV-201 is a cell therapy produced by MAT that consists of the participant's autologous CD34+ hematopoietic stem and progenitor cells (HSPCs) enriched with allogeneic placental-derived mitochondria, manufactured in Minovia's GMP facility.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants aged from 18 years old and above.
2. Low Risk MDS diagnosis with R-IPSS score of ≤3 with mutational burden and/or low burden of high-risk mutations as defined by IPSS-M.
3. Participant has anemia and is blood transfusion dependent (received 2 or more units of packed blood per /4 weeks for at least 8 weeks before enrollment).
4. A baseline natural history of the participant is available, including anemia and transfusions frequency at least 6 months before enrollment.
5. Participant has utilized all existing treatments for low risk MDS that are approved and available to him or is not medically eligible for those treatment options.
6. Participant is not eligible for Allogeneic Bone Marrow Transplantation.
7. Participant is medically able to undergo the study interventions, as determined by the investigator.
8. Participant and/or legal guardian(s) able to understand and provide voluntary written informed consent.

Exclusion criteria:

1. History of infection with HIV-1, HIV-2, or HTLV I/II.
2. Current active infection with HBV , HCV, HTLV I/II, Treponema Pallidum or HIV I-II.
3. Participant is unable to undergo apheresis.
4. Participant has known hypersensitivity to murine proteins or iron-dextran.
5. Participant has chronic severe infection.
6. Participant has disease or condition that may risk the participant or interfere with the ability to interpret the study results.
7. History of treatment for malignant disease (other than excision of non-melanoma skin cancer) in the last 2 years
8. Pregnancy or breastfeeding
9. History of treatment with gene therapy, bone marrow or allogeneic cord blood transplantation.
10. Currently participating in another clinical trial, or participation in another clinical trial within 1 year prior to study enrollment.
11. In the opinion of the Investigator, the participant is unsuitable for participating in the study for any reason.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-05-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-related adverse events | 1 year
  Occurrence of treatment-related adverse events as assessed by CTCAE v5.0 following MNV-201 infusion, during a follow up period of 12 months following first dosing (Part 1) and 6 months following second dosing (Part 2), where relevant.

SECONDARY OUTCOMES:
Anemia assessment | 1 year
  Hemoglobin rise measured by CBC of at least 1 g/dL from baseline during a follow up period of 6- and 12-months post treatment (Part 1) or 6 months post
Blood transfusion assessment | 1 year
  Reduction in frequency of blood transfusions during a follow up period of 6- and 12-months post treatment (Part 1) or 6 months post treatment (Part 2) compared to the 6 months period before treatment.
Assessment of Quality of Life by the Functional Assessment of Cancer Therapy - Anemia | 1 year
  Change in health-related quality-of-life (HRQoL) assessed by the Functional Assessment of Cancer Therapy - Anemia (FACT-An) from baseline during a follow up period of 6- and 12-months post treatment (Part 1) or 6 months post treatment (Part 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel, Israel

IPD SHARING:
Plan to Share IPD: No